CLINICAL TRIAL: NCT01170897
Title: A Phase 1, Multicenter, Open-Label, Dose-Escalation, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of PEGPH20 With Initial Dexamethasone Premedication Given Intravenously to Patients With Advanced Solid Tumors
Brief Title: Study of PEGPH20 With Initial Dexamethasone Premedication Given Intravenously to Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: HALO-109-102
Record Dates: First submitted 2010-07-26; First posted 2010-07-27 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2012-09

CONDITIONS: Solid Tumor
Keywords: PEGPH20; PEGylated Recombinant Human Hyaluronidase; Metastatic or Locally Advanced Solid Tumors
MeSH Terms: conditions — Neoplasm Metastasis | interventions — PEGPH20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Maximally Tolerated Dose (Other): To identify the maximally tolerated dose (MTD) of PEGPH20.
  Interventions: Drug: PEGPH20

INTERVENTIONS:
Drug: PEGPH20 — PEGylated Recombinant Human Hyaluronidase

SUMMARY:
This is an open-label, multicenter, dose-escalation, safety, tolerability, pharmacokinetic and pharmacodynamic study in patients with advanced solid tumors.

DETAILED DESCRIPTION:
A study of PEGylated recombinant human hyaluronidase (PEGPH20) administered on a twice weekly schedule for 28 days followed by a weekly dosing schedule in patients with advanced solid tumors who have either failed to respond to standard therapy or for whom no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed, IRB-approved informed consent form.
* Pathologic (histologic or cytologic) confirmation of metastatic or locally advanced solid tumor.
* Patients must have a pathologically documented, definitively diagnosed, advanced solid tumor that is refractory to standard treatment, for which no standard therapy is available or the patient refuses standard therapy.
* One or more tumors measurable by RECIST criteria.
* Karnofsky performance status ≥ 70%.
* Ejection fraction ≥ 50%, determined by echocardiogram.
* Life expectancy at least 3 months.
* Age ≥ 18 years.
* Acceptable organ function; normal hepatic, renal and hematopoietic function.
* Negative serum or urine pregnancy test result in women of childbearing potential.

Exclusion Criteria:

* Known brain metastasis.
* New York Heart Association Class III or IV cardiac disease, myocardial infarction within 6 months of enrollment, or cardiac arrhythmia requiring medical therapy.
* Active, uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
* Patients with uncontrolled diabetes (requiring medication change within 30 days of screening), or requiring insulin therapy.
* Heparin therapy.
* Known infection with HIV, hepatitis B, or hepatitis C.
* Known allergy to hyaluronidase.
* Women currently breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximally Tolerated Dose (MTD) of PEGPH20 when given to patients with cancer | To be evaluable for MTD determination, a patient must have completed the Cycle 1 study drug doses and the associated assessments for safety and toxicity evaluation
  The PEGPH20 monotherapy MTD is the highest dose at which no more than one of six evaluable patients experience Dose-Limiting Toxicity (DLT)
Safety endpoints including assessment of both serious and non-serious AEs | From Day 1 of Treatment Cycle 1, thru to Follow-up (within 28 days after last dose of PEGPH20)
  All safety data will be evaluated using the NCI CTCAE scoring system (version 4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Joy Zhu, M.D., Study Director — Halozyme Therapeutics
Locations (5):
- United States (5):
  - Ramesh K. Ramanathan M.D., Scottsdale, Arizona
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - cCare - California Cancer Associatesfor Research Excellence, Encinitas, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Jeffrey R. Infante, Nashville, Tennessee